CLINICAL TRIAL: NCT03698175
Title: Can Brief Daily Mental Exercises Change the Way the Human Brain Processes Certain Kinds of Information?
Brief Title: Effects of a Brief Mental Exercise on Emotional Processing
Acronym: BME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MS IDREC R49254
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Emotional Processing; Mental Exercise
Keywords: Emotion; Cognition; Positive psychology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three good things exercise (Experimental)
  Interventions: Behavioral: Three good things exercise
- Unspecific childhood memory recall exercise (Placebo Comparator)
  Interventions: Behavioral: Placebo exercise

INTERVENTIONS:
Behavioral: Three good things exercise — Participants are asked to remember each evening three things that went well during their day and to write them down in a journal including a short explanation of why they think each of them has happened.
  Arms: Three good things exercise
Behavioral: Placebo exercise — Participants are asked to briefly recall a childhood memory (no further specification) and to write it down including a short explanation why they think it has happened.
  Arms: Unspecific childhood memory recall exercise

SUMMARY:
The aim of this study is to explore whether a brief mental exercise (developed and widely advocated in the field of positive psychology) can change the processing of emotion-related information in a similar way as previously observed for antidepressant drugs. Healthy volunteers are randomly allocated to a 7-day practice of the "Three Good Things" (TGT) exercise or a previously used placebo exercise (unspecified childhood memory recall) with study participants as well as investigators being blind as to which practice is conducted. After a 7-day practice period, all study participants undergo testing with the Oxford Emotional Test Battery, an established battery of cognitive tasks that allow to assess how emotional information is processed. The working hypothesis of the study is that the TGT exercise, as compared to the placebo exercise, can push the processing of emotional information towards a prioritisation of positive (relative to negative) input.

DETAILED DESCRIPTION:
Background and objective:

Previous research indicates that various physiological treatments for depression (especially antidepressant drugs) can induce positive biases in emotional information processing and it has been suggested that this might be a crucial common mechanism through which they exert their clinical effects. This study aims to investigate whether similar positive biases can also be induced by a brief mental exercise (developed and widely used within the field of positive psychology) that has previously been shown to have antidepressant and/or happiness-enhancing effects.

Methods:

Using a double-blind, parallel-group design, 100 healthy volunteers (male and female) are randomly allocated to a 7-day mental exercise practice conducting either the widely reported Three Good Things (TGT) exercise or a previously established placebo condition (unspecific childhood memory recall). After 7 days of practice, all participants undergo testing with the Oxford Emotional Test Battery in order to assess emotional information processing in different cognitive domains. This battery consists of a facial expression recognition task, an emotional categorization task, an emotional dot probe task, an emotional recall task and an emotional recognition task. In addition, prior to and immediately after the 7-day practice period salivary cortisol awakening response and subjective state (using various questionnaires) is assessed.

Hypotheses:

The working hypothesis of the study is that, similar to physiological antidepressant interventions, the TGT exercise (as compared to the placebo exercise) might induce biases towards positive stimuli in multiple cognitive domains.

Implications of the study:

This study will show whether engaging in a simple mental exercise can alter emotional information processing in a similar way as previously observed for antidepressant drugs and other physiological interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male
2. Age: 18 to 65 years
3. Good general health
4. Competency to give informed consent

Exclusion Criteria:

1. Any current or past psychiatric disorder
2. Any first-degree relative with a diagnosis of schizophrenia-spectrum or other psychotic disorder, bipolar disorder, or depressive disorder
3. Regular engagement in mental exercises specifically aimed at improving cognitive abilities (concentration, attention, memory etc.), mood, or general well-being, such as (online) cognitive training, positive psychology exercises, regular meditation or mindfulness practices, yoga practices, or psychotherapeutic exercises.
4. Regular engagement in any of the exercises outlined above within the last 6 months.
5. Any severe medical condition not stabilized at the time of the study (e.g. asthma, heart disease, epilepsy)
6. Any current or past physical illness that has the potential to significantly affect mental functioning (e.g. stroke, Parkinson's disease, multiple sclerosis)
7. Current intake of medication that has a significant potential to affect mental functioning, or intake of such medication in the previous 3 months (e.g. antidepressants, neuroleptics, tranquilizers)
8. Any intake of recreational drugs in the last 3 months before the experiment
9. Regular consumption of higher doses of alcohol (more than 2 pints of beer or equivalent on more than 3 days a week within the last month)
10. Any other reasons that preclude participants from full participation in the experiment (e.g. insufficient knowledge of English language)
11. Any other condition which can make participation in the study harmful for a participant, or which can severely compromise the quality of the data (e.g. low intellectual functioning)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Performance in a facial expression recognition task | Completed at day 8 after exercise has been started
  Participants are presented with individual pictures of facial expressions of emotions. Each presented face displays one of six basic emotions (anger, disgust, fear, happiness, sadness, or surprise). Each emotional expression is presented at different levels of intensity which have been created by combining shape and texture features of the two extremes "neutral" (0%) and "full prototypical emotion" (100%) to varying degrees. Examples of neutral facial expressions are presented as well. Participants are instructed to correctly classify each facial expression as angry, disgusted, fearful, happy, sad, surprised or neutral both as quickly and as accurately as possible. Responses are made by pushing one out of seven labelled keys on a response box. Hit rates, false alarm rates, and reaction times for correct classifications are measured separately for each emotion.

SECONDARY OUTCOMES:
Performance in an emotional categorisation task | Completed at day 8 after exercise has been started
  Participants are presented with positive and negative personality descriptors and are asked to classify the valence of each word. These words describe either extremely agreeable/positive characteristics (e.g. "cheerful", "honest", "optimistic") or extremely disagreeable/negative characteristics (e.g. "domineering", "untidy", "hostile") and are presented individually in the centre of the screen. Participants are instructed to imagine themselves overhearing someone describing them with each of the words and to indicate as quickly and accurately as possible whether they would like or dislike to be described with each of the words. Responses are made by pressing a correspondingly labelled key on a button box. Reaction times for correct classifications are measured separately for positive and negative words.
Performance in an emotional faces dot probe task | Completed at day 8 after exercise has been started
  Pictures of positive and negative emotional stimuli (happy and fearful facial expressions) are presented individually together with a matched neutral stimulus (neutral face). On each trial, one stimulus is shown above and the other below a central fixation point. Subsequently, a probe appears behind one of the stimuli and participants have to correctly classify the probe as quickly and as accurately as possible. Stimuli can be masked (i.e. presented very briefly and followed by a jumbled face) or unmasked (i.e. presented for a longer period without a subsequent masking stimulus). Reaction times for correct responses are recorded and vigilance scores are calculated for masked and unmasked positive and negative stimuli by subtracting reaction time data from trials when the probe appeared in the same position as the emotional stimulus (congruent trials) from trials when the probe appeared in the opposite position to the emotional stimulus (incongruent trials).
Performance in an emotional recall task | Completed at day 8 after exercise has been started
  Following a delay period after the emotional categorisation task (about 15 min), emotional recall memory is assessed. Participants are asked to recall and write down as many words as possible from the emotional categorization task. Numbers of correctly and incorrectly recalled positive and negative words are measured.
Performance in an emotional recognition task | Completed at day 8 after exercise has been started
  Following the emotional recall task, emotional recognition memory is assessed by presenting participants with the original personality descriptors plus an equal number of matched distractor words (50% positive, 50% negative). Participants are asked to indicate for each word as accurately and as quickly as possible whether they recognise it from the emotional categorization task. Numbers of correctly and incorrectly recognised items as well as reaction times for correct recognitions are measured separately for positive and negative words.
Change in cortisol awakening response | Completed at day 8 after exercise has been started
  Salivary cortisol is assessed prior to and after completion of the 7-day exercise period. For each assessment, participants have to provide five saliva samples taken in their own home (0, 15, 30, 45, and 60 minutes after awakening).

OTHER OUTCOMES:
Change in subclinical depressive symptoms | Completed at day 8 after exercise has been started
  Center for Epidemiologic Studies Depression Scale Revised. Standard questionnaire to assess symptoms of depression. Total score ranging from 0 to 60 with higher scores indicating higher levels of depressive symptoms.
Change in authentic happiness | Completed at day 8 after exercise has been started
  Authentic Happiness Inventory. Questionnaire developed to assess authentic happiness levels. Scores ranging from 0 to 120 with higher scores indicating higher happiness levels.
Change in subjective anxiety | Completed at day 8 after exercise has been started
  State-Trait Anxiety Inventory. Standard questionnaire for subjectively felt anxiety. Two scores: (1) State anxiety: ranging from 20 to 80 (higher scores indicating higher state anxiety levels). (2) Trait Anxiety: ranging from 20 to 80 (higher scores indicating higher trait anxiety levels).
Change in subjective mood and energy | Completed at day 8 after exercise has been started
  Zersen's Befindlichkeits-Skala. Standard questionnaire for subjectively felt mood and energy levels. Total score ranging from 0 to 112. Subscores: Mood (ranging from 0 to 94) and Energy (ranging from 0 to 18). Sum of subscores for mood and energy provide total score. Higher scores represent worse subjective mood and energy
Change in positive and negative affect | Completed at day 8 after exercise has been started
  Positive and Negative Affect Schedule. Standard questionnaire for subjectively felt positive and negative affect. Two scores: (1) Positive score: ranging from 10 to 50 (higher score representing greater extent of positive affect). (2) Negative score: ranging from 10 to 50 (higher score representing greater extent of negative affect).
Change in subclinical depressive symptoms | Completed at day 8 after exercise has been started
  Beck Depression Inventory. Standard questionnaire for assessment of depression severity. Scores ranging from 0 to 63 with higher scores indicating greater depressive severity.
Change in subjective state | Completed at day 8 after exercise has been started
  Visual Analogue Scales of different subjective states (anxious, alert, happy, sad, angry, disgusted, afraid). Minimum = 0 mm ("Not at all") , Maximum = 96 mm ("Extremely"). Greater scores represent greater extent of felt emotions.
Type of recorded positive events | Completed at day 8 after exercise has been started
  Written records of positive events will be coded according to theme. Prevalence of each theme will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom